CLINICAL TRIAL: NCT00395187
Title: A Small Clinical Study: Photodynamic Therapy to Treat Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10514
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Photodynamic Therapy

SUMMARY:
This study will investigate the efficacy of Photodynamic Therapy (PDT), which is the therapeutic use of photochemical reactions, in treating hidradenitis suppurativa (HS), a chronic inflammatory condition affecting areas of skin with sweat glands. We expect that PDT is effective in treating HS.

DETAILED DESCRIPTION:
This study will investigate the efficacy of PDT using aminolevulinic acid (ALA) and either blue light or intense pulsed light on active lesions of HS. We will attempt to validate the success noted in a previously published case series using PDT with ALA and blue light (Gold, Bridges et al). We will evaluate effect of treatment by number of lesions, global disease severity, and patient self-assessment with the Dermatology Life Quality Index (DLQI).

Detailed informed consent will be obtained prior to treatment at study enrollment. The first four treatment visits will involve clinical evaluation, photography and application of the ALA to the affected area. After a 45 minute incubation period, the area will be washed and then treated with either blue light or intense pulsed light (IPL), depending on body area/investigator choice. One and three-month follow-up visits will involve evaluation of efficacy, but no active treatment.

Gold M, Bridges TM, et al. ALA-PDT and blue light therapy for hidradenitis suppurative. J Drugs Dermatol. 2004; 3 (1 Suppl):S32-5.

ELIGIBILITY:
Inclusion Criteria:

* multiple lesions consistent with HS in axillae/groin
* history of no or poor response to at least one treatment modality
* no active treatment in the 2 weeks prior to study initiation

Exclusion Criteria:

* Pregnancy/lactation
* photosensitizing drug use within 30 days of start of study
* active infection needing antibiotics
* history of porphyria or photosensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Active and inactive lesion count | 0,1,2,3,4,8,16 weeks

SECONDARY OUTCOMES:
Regional disease severity will be assessed at each visit. Global Severity Score will be assigned by investigator. Assessed at all 6 visits, Patient self -assessment (DLQI) at visits 4-6,-Digital photographs-all 6 visits,Safety/adverse event monitoring. | 0,1,2,3,4,8,16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Aires, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States